CLINICAL TRIAL: NCT07403474
Title: Combined Use of a Respiratory Multiplex PCR and Algorithm-based Therapy to Improve Early Optimization of Antibiotic Therapy in Critically Ill Patients With Ventilator-associated Pneumonia : a Bicentric, Parallel-group, Randomized Controlled Trial.
Brief Title: Combined Use of a Respiratory Multiplex PCR and Algorithm-based Therapy to Improve Early Optimization of Antibiotic Therapy in Critically Ill Patients With Ventilator-associated Pneumonia
Acronym: SMART-VAP
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-A02343-46
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Ventilator Associated Pneumonia ( VAP)
Keywords: mPCR; ventilator associated pneumonia; algorithm-based therapy
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Intervention Model Description: This prospective, randomized, controlled, blinded, parallel-group study evaluates a semi-guided antibiotic strategy based on respiratory mPCR integrated with a locally derived decision algorithm, compared with standard antibiotic care in intensive care patients with ventilator-associated or nosocomial pneumonia.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors (investigator-delegated evaluators, different from those who performed the procedure) will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combined use of mPCR and algorithm-based therapy (Experimental): strategy combining respiratory mPCR on a deep respiratory sample obtained by mini bronchoalveolar lavage and algorithm-based therapy developed using local epidemiology
  Interventions: Procedure: strategy combining respiratory mPCR and algorithm-based therapy developed using local epidemiology
- Conventional strategy for antibiotic therapy at discretion of ICU physicians (No Intervention): The conventional strategy is based on the clinician's choice in accordance with best practice recommendations, without the combined use of respiratory mPCR and algorithm-based therapy.

INTERVENTIONS:
Procedure: strategy combining respiratory mPCR and algorithm-based therapy developed using local epidemiology — strategy combining respiratory mPCR carried out either by mini bronchoalveolar lavage (BAL) via bronchoscopy or by blind mini BAL, and algorithm-based therapy developed using local epidemiology for the early optimization of initial antibiotic therapy
  Arms: combined use of mPCR and algorithm-based therapy

SUMMARY:
Assess the impact of a strategy combining respiratory mPCR and algorithm-based therapy developed using local epidemiology on the early optimization of initial antibiotic therapy for ventilator-associated pneumonia (VAP) (intervention), compared to a conventional strategy (control).

A bicentric, parallel-group, randomized controlled trial. The primary assessment criterion is the proportion of early optimized antibiotic therapy within 24 hours of respiratory sampling.

DETAILED DESCRIPTION:
In both arms, for eligible patients with VAP, a deep respiratory sample collection is performed prior to inclusion. This collection is carried out either by mini bronchoalveolar lavage (BAL) via bronchoscopy or by blind mini BAL in alignment with the protocolized procedure. Initial antibiotic therapy is initiated after the deep sample has been taken according to the discretion of the attending clinician and in accordance with good practice recommendations. Both groups have their samples analyzed using conventional techniques. First, there is a direct examination, followed by culture and susceptibility testing, which is used as the gold standard technique for evaluating the primary endpoint.

In the intervention arm, in addition to conventional techniques, a broad-panel respiratory mPCR is performed before the 12th hour following achievement of the deep respiratory sample on the collected BAL. Once the mPCR results are received, the clinician adjusts the initial antibiotic therapy using algorithm-based therapy developed using local epidemiology in order to optimize treatment as early as possible.

In the control arm, the strategy is based on the clinician's choice in accordance with best practice recommendations without the combined use of respiratory mPCR and algorithm-based therapy. The deep respiratory sample is analyzed using conventional methods. Initial antibiotic treatment is therefore adapted by the clinician in charge of the patient according to departmental practices based on best practice recommendations, taking into account the results of the direct examination, culture, and susceptibility testing.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with VAP (mechanical ventilation and hospitalization ≥ 48 hours) and deep respiratory sample by mini BAL < 12 hours. The diagnosis of pneumonia includes two clinical criteria among fever (≥38.3°C), purulent sputum or aspiration, hyperleukocytosis (>12,000 WBC/mm³) or leukopenia (<4,000 WBC/mm³), hypoxemia, auscultatory signs in the affected area, and a newly-appeared parenchymal infiltrate
* Patient receiving initial probabilistic antibiotic therapy for VAP suspicion
* Informed consent or emergency procedure
* Patient affiliated with or beneficiary of a health insurance plan.

Non inclusion Criteria:

* Pregnancy
* Congenital immunodeficiency;
* HIV infection with the lymphocyte CD4 count below 200/mm3 or unknown in the last year;
* Acute hematologic malignancy;
* Neutropenia (<1 leucocyte/mL or < 0.5 neutrophil/mL);
* Immunosuppressive drugs within the previous 30 days, including anti-cancer - Chemotherapy and anti-rejection drugs for organ/bone marrow transplant
* Corticosteroids ≥ 20 mg/d of prednisone equivalent for more than 14 days
* Known allergy to beta-lactams
* Moribund patient or death expected from underlying disease during the current admission;
* Patient deprived of liberty or under legal protection measure;
* Participation in another interventional trial.

Exclusion criteria :

* mPCR non available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of a combined use a broad panel respiratory mPCR and an algorithm-based therapy developed using local epidemiology on the early optimization of initial antibiotic therapy for VAP, as compared to a conventional strategy | Day 1
  Proportion of patients receiving optimized antibiotic therapy defined as effective antibiotic therapy and for which antibiotic de-escalation, when recommended, was performed early, within 24 hours after deep respiratory sampling.

SECONDARY OUTCOMES:
Duration of exposure to broad-spectrum antibiotic therapy. | Day 28
  Average number of days of broad-spectrum antibiotic administration per patient at day 28
Compare expected and actual time frames for optimizing antibiotic therapy in the two arms. | day 28
  Time in hours between deep respiratory sampling and optimization of antibiotic therapy.
Quantify early antibiotic de-escalation in the two groups under study | day 1 and day 7
  Early and broad-spectrum antibiotic sparing according to the modified Antibiotic Spectrum Index (ASIm) de-escalation score (from No antibiotics (0) to very broad (≥8))
Rate of Clinical Cure at Day | day 7
  use test of cure at day 7
Mechanical ventilation at day 28 | day 28
  mechanical ventilation free-days at day 28
lenght of stay in ICU at day 28 | day 28
  ICU free-days at day 28
Number of organ-failure free days (based on SOFA) at day 28 | day 28
  Number of organ-failure free days (based on SOFA) at day 28
Mortality at day 28 | day 28
  Mortality at 28
Sensitivity, specificity, and likelihood ratios of the broad panel mPCR Film Array for the diagnosis of pneumonia, taking the conventional microbiological tests as reference | day 28
  Sensitivity, specificity, and likelihood ratios of the broad panel mPCR Film Array for the diagnosis of pneumonia, taking the conventional microbiological tests as reference
Incidence rates of infection or colonization with multidrug resistant bacteria and Clostridium difficile infections at day 28 | day 28
  Incidence rates of infection or colonization with multidrug resistant bacteria and Clostridium difficile infections at day 28
Cost of the total hospital admissions | day 28
  Total Hospitalization Cost per Participant at Day 28 (Including ICU Stay, Antimicrobial Therapy, Microbiological Diagnostic Workup, and Infection Relapse Costs)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nîmes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No